

### **Clinical Research Protocol**

# Trapezio – metacarpal arthroplasty: comparison of ARPE® prosthesis with the literature

PROTOCOL NUMBER (Study ID): ORTHO.CR.E16

PROTOCOL VERSION: V1.0 dd 12 Nov 2012

**GENERAL INFORMATION** 

Study Sponsor: BIOMET Global Supply Chain Center B.V.

Toermalijnring 600 3316 LC Dordrecht The Netherlands



## **Clinical Research Protocol**

| TITLE | Trapezio-metarcarpal arthroplasty: a comparison of ARPE prosthesis with the literature |
|---|---|
| SHORT TITLE | Arpe prospective study |
| DESIGN | Non-controlled, prospective cohort study in single centre |
| STUDY<br>DURATION | 2013- 2020 |
| STUDY CENTRE | Single centre in Belgium |
| POPULATION | Inclusion of 100 subjects at single centre |
| PRIMARY<br>Research<br>objectives | The primary objective is to compare functional outcome at 3 years after trapezio-metarcarpal arthroplasty with trapeziectomy and trapeziectomy with ligament reconstruction and tendon interposition. Literature values obtained by a recently published meta analysis¹ will be used. |
| SECONDARY<br>Research<br>Objectives | Secondary objectives are: - to compare functional outcome at 1 and at 5 years after trapezio-metarcarpal arthroplasty with trapeziectomy and trapeziectomy with ligament reconstruction and tendon interposition - to determine pre- and postop HR QOL - Incidence of RLL at each f/up time point. Literature values from the same meta analysis¹ will be used. |
| OUTCOME<br>Measures | Patients will be assessed at preoperatively, and at 1, 3 and 5 years postoperatively. Outcomes as described by Li et al <sup>1</sup> will be measured: grip strength, tip pinch strength, key pinch strength, pain, occurrence of adverse events, hand function. |
| Follow-up time | Patients will be part of a longitudinal follow-up program with follow-ups at 1, 3, 5 years. |
| Enrollment time | 2 Years |

Study: Arpe prospective study



#### **Clinical Research Protocol**

#### **STATISTICS**

#### SAMPLE SIZE CALCULATION

Based on a publication from Davis et al<sup>2</sup> we expect the standard deviation in the study population for key pinch, tip pinch, and grip strength to be 0.82, 1.65 and 10.3, respectively. Setting alpha at 0.05 and beta at 0.10, and assuming a MIREDIF (Minimally Relevant Difference) of 0.5 x Standard Deviation, an attrition rate of 10%, and data to be approximately normally distributed, the required sample size will be 96 ( $\approx$  100) subjects.

#### STATISTICAL PROTOCOL

Continuous variables (e.g. age) will be summarized using the mean and standard deviation (SD). If the distribution of measurements is asymmetrical, the median and the interquartile range will be provided. For ordinal and nominal data proportions should be employed. Inferential statistics will be based on the unpaired t-test, or the Mann-Whitney test, depending on normality of the data.

#### **REFERENCES**

- 1. LI YK, WHITE C, IGNACY TA, THOMA A. COMPARISON OF TRAPEZIECTOMY AND TRAPEZIECTOMY WITH LIGAMENT RECONSTRUCTION AND TENDON INTERPOSITION: A SYSTEMATIC LITERATURE REVIEW. PLASTIC AND RECONSTRUCTIVE SURGERY. 2011 JUL;128(1):199-207. PUBMED PMID: 2139956
- 2. DAVIS TR, PACE A. TRAPEZIECTOMY FOR TRAPEZIOMETACARPAL JOINT OSTEOARTHRITIS: IS LIGAMENT RECONSTRUCTION AND TEMPORARY STABILISATION OF THE PSEUDARTHROSIS WITH A KIRSCHNER WIRE IMPORTANT? THE JOURNAL OF HAND SURGERY, EUROPEAN VOLUME. 2009 JUN;34(3):312-21. PUBMED PMID: 19321528.